CLINICAL TRIAL: NCT00779753
Title: Determination of Lysine Requirement in the Parenterally Fed Neonate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Karen Chapman, Clinical Research Nurse Specialist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0019880597
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Parenteral Lysine Requirements; Parenteral Feedings
Keywords: Parenteral Feeding; Neonate; Lysine
MeSH Terms: interventions — amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neonates (Experimental): Sixteen neonates admitted to the Neonatal Intensive Care Unit (NICU) at the Hospital for Sick Children (SickKids) will be required for this study. The diagnoses will include, but are not limited to, the following: Trachea-esophageal fistula and/or esophageal atresia, Congenital diaphragmatic hernia, imperforate anus, Hirschsprung's disease, Malrotation with or without volvulus, Intestinal atresias, Gastroschisis, Omphalocele, Necrotizing enterocolitis, Respiratory distress syndrome.
  Interventions: Dietary Supplement: Amino Acid Solution with different amount of Lysine

INTERVENTIONS:
Dietary Supplement: Amino Acid Solution with different amount of Lysine — The infants will be placed on a standard Primene solution for the first 24 hours of the study to obtain baseline values. During the second 24 hours they will receive an amino acid solution that has a different amount of lysine currently found in Primene, all lipid, CHO, minerals, vitamins and trace elements will remain unchanged. The Parenteral lysine will be studied at the following intake levels: 100, 110, 120, 130, 135, 140, 145, 150 , 155, 165, 170, 180, 200, 230, 245, 260mg/kg/d. The minimum energy intake will be 85-90 kcal/kg/day.
  Other Names: Trophamine; Primene

SUMMARY:
The purpose of this study is to establish the parenteral lysine requirements for neonates.

DETAILED DESCRIPTION:
It is important to identify the appropriate level of lysine requirements for parenterally fed neonates as this amino acid is the limiting amino acid in the diet of neonates. Feeding lysine at requirement improves the likelihood that other amino acids will be utilized appropriately for building proteins. In addition, lysine plays a major role in calcium absorption, development of muscle proteins and in the production of hormones, enzymes and antibodies. We believe that the lysine requirement will be 158 mg/kg/day which is significantly lower than the current 267 and 327 mg/kg/d that is found in the current Trophamine and Primene parenteral solutions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable neonates on TPN
* minimum of 2.5 g/kg/d protein and 85 - 90 kcal/kg/d)
* Post conception age of ≥ 34 weeks gestation and appropriate for gestational age
* Weight of ≥ 1.5 kg
* NPO or ≤10% of total protein requirement consumed enterally

Exclusion Criteria:

* Infants on mechanical ventilators, supplemental oxygen or who are receiving medications that would alter protein or energy metabolism (ie. corticosteroid therapy, etc)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Oxydation of the Indicator Amino Acid L-[1-13C] phenylalanine will be measured through urine samples to determine urinary phenylalanine enrichment | 2 days

SECONDARY OUTCOMES:
Breath samples will be collected for the measurement of CO2 enrichment in expired air | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chapman, RN, PhD (c), Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chapman KP, Elango R, Ball RO, Pencharz PB. Splanchnic first pass disappearance of threonine and lysine do not differ in healthy men in the fed state. J Nutr. 2013 Mar;143(3):290-4. doi: 10.3945/jn.112.168328. Epub 2013 Jan 16. PMID 23325919
- [Derived] Chapman KP, Courtney-Martin G, Moore AM, Langer JC, Tomlinson C, Ball RO, Pencharz PB. Lysine requirement in parenterally fed postsurgical human neonates. Am J Clin Nutr. 2010 Apr;91(4):958-65. doi: 10.3945/ajcn.2009.28729. Epub 2010 Feb 17. PMID 20164307